CLINICAL TRIAL: NCT03548337
Title: A PHASE 4, RANDOMIZED, OPEN-LABEL TRIAL TO DESCRIBE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF 13- VALENT PNEUMOCOCCAL CONJUGATE VACCINE FORMULATED IN MULTIDOSE VIALS WHEN GIVEN WITH ROUTINE PEDIATRIC VACCINES IN HEALTHY INFANTS IN INDIA
Brief Title: Study To Describe The Safety, Tolerability, And Immunogenicity Of 13- Valent Pneumococcal Conjugate Vaccine Formulated In Multidose Vials When Given With Routine Pediatric Vaccines In Healthy Infants In India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B4671004; INDIA INFANT MDV (Other: Alias Study Number); 2016-005134-29 (EudraCT Number)
Record Dates: First submitted 2018-05-22; First posted 2018-06-07 (Actual); Results first posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 13vPnC with 2-PE from a MDV (Active Comparator): Multi Dose Vial with preservative
  Interventions: Biological: 13vPnC
- 13vPnC without 2-PE in a PFS (Active Comparator): Pre Filled Syringe without preservative
  Interventions: Biological: 13vPnC

INTERVENTIONS:
Biological: 13vPnC — 13vPnC MultiDose Vial with preservative compared to a Prefilled syringe containing 13vPnC without any preservative

SUMMARY:
A Phase 4 Study To Describe The Safety, Tolerability, And Immunogenicity Of 13- Valent Pneumococcal Conjugate Vaccine Formulated In Multidose Vials When Given With Routine Pediatric Vaccines In Healthy Infants In India

DETAILED DESCRIPTION:
A Phase 4, Randomized, Open-label Trial To Describe The Safety, Tolerability, And Immunogenicity Of 13- Valent Pneumococcal Conjugate Vaccine Formulated In Multidose Vials When Given With Routine Pediatric Vaccines In Healthy Infants In India

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the parent(s)/legal guardian(s) has/have been informed of all pertinent aspects of the study.
2. Parent(s)/legal guardian(s)/caregiver(s) willing and able to comply with scheduled visits, treatment plan, and other study procedures.
3. Aged 6 weeks (42 to 72 days) at the time of vaccination. (The day of birth is considered Day 0.)
4. Available for the entire study period and whose parent(s)/legal guardian(s)/caregiver(s) can be reached by telephone.
5. Healthy infant as determined by medical history, physical examination, and judgment of the investigator.
6. Weight of 3.0 kg or greater at the time of vaccination.

Exclusion Criteria:

1. Infant who is a direct descendant (child, grandchild) of

   * Investigator site staff members directly involved in the conduct of the study, or
   * Site staff members otherwise supervised by the investigator, or
   * Pfizer employees directly involved in the conduct of the study.
2. Participation in other studies involving investigational drug(s) within 28 days prior to study entry and/or during study participation. Participation in purely observational studies is acceptable.
3. Previous vaccination with licensed or investigational pneumococcal conjugate vaccine.
4. A previous anaphylactic reaction to any vaccine or vaccine-related component.
5. Contraindication to vaccination with pneumococcal conjugate vaccine, or any other vaccine or vaccine component. Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
6. Known or suspected immune deficiency or suppression, including known human immunodeficiency virus infection.
7. Major known congenital malformation or serious chronic disorder.
8. Significant neurological disorder or history of seizure including febrile seizure, or significant stable or evolving disorders such as cerebral palsy, encephalopathy, hydrocephalus, or other significant disorders. Does not include resolving syndromes due to birth trauma such as Erb's palsy.
9. Other acute or chronic medical condition including recent laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
10. Receipt of blood products or gamma globulin (including hepatitis B immunoglobulin and monoclonal antibodies, eg, Synagis).

Ages: 42 Days to 72 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 301 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- India (7):
  - B. J. Medical College & Civil Hospital, Ahmedabad, Gujarat
  - Manipal Hospital, Bengaluru, Karnataka
  - KEM Hospital Research Centre, Pune, Maharashtra
  - Bharati Vidyapeeth University Medical College, Pune, Maharashtra
  - Sri Ramachandra Hospital, Chennai, Tamil Nadu
  - Kanchi Kamakoti Childs Trust Hospital, Chennai, Tamil Nadu
  - Sir Ganga Ram Hospital, New Delhi

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Lalwani SK, Ramanan PV, Sapru A, Sundaram B, Shah BH, Kaul D, Karthik Nagesh N, Kalina WV, Chand R, Ding M, Suroju S, Scott DA, Lockhart SP. Safety and immunogenicity of a multidose vial formulation of 13-valent pneumococcal conjugate vaccine administered with routine pediatric vaccines in healthy infants in India: A phase 4, randomized, open-label study. Vaccine. 2021 Nov 5;39(46):6787-6795. doi: 10.1016/j.vaccine.2021.09.029. Epub 2021 Oct 14. PMID 34656378
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B4671004

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC: Multi-dose Vial (With Preservative): Infant series: participants were randomized to receive a single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) with preservative 2-phenoxyethanol (2-PE) from a multi-dose vial (MDV), intramuscularly at age of 6 weeks (Vaccination 1), 10 weeks (Vaccination 2) and 14 weeks (Vaccination 3) along with 2 routine vaccines: 1) diphtheria, tetanus, and pertussis; Haemophilus influenzae type b; and hepatitis B virus (DTP-Hib-HBV) vaccine, 2) rotavirus vaccine. Participants were followed-up to 1 month after Vaccination 3. Infant series was followed by toddler dose. Toddler dose: participants were administered with a single 0.5 mL dose of 13vPnC vaccine with preservative 2-PE from MDV, intramuscularly at age of 12 months (Vaccination 4) along with routine hepatitis A virus vaccine. Participants were followed-up to 1 month after Vaccination 4. Different limbs were used to administer study vaccine and routine vaccines (according to local clinical practice).
- 13vPnC: Single-dose Prefilled Syringe (Without Preservative): Infant series: participants were randomized to receive a single 0.5 mL dose of 13vPnC without preservative 2-PE from a single-dose prefilled syringe (PFS), intramuscularly at age of 6 weeks (Vaccination 1), 10 weeks (Vaccination 2) and 14 weeks (Vaccination 3) along with 2 routine vaccines: 1) DTP-Hib-HBV vaccine, 2) rotavirus vaccine. Participants were followed-up to 1 month after Vaccination 3. Infant series was followed by toddler dose. Toddler dose: participants were administered with a single 0.5 mL dose of 13vPnC vaccine without preservative 2-PE from single dose PFS, intramuscularly at age of 12 months (Vaccination 4) along with routine hepatitis A virus vaccine. Participants were followed-up to 1 month after Vaccination 4. Different limbs were used to administer study vaccine and routine vaccines (according to local clinical practice).
Period: Infant Series
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Started | 151 | 150
Vaccination 1 | 150 | 150
Vaccination 2 | 144 | 144
Vaccination 3 | 144 | 141
Completed | 139 | 139
Not Completed | 12 | 11
Not completed — Withdrawal by Parent/Guardian | 8 | 8
Not completed — No Longer Met Eligibility Criteria | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Randomized but Not Vaccinated | 1 | 0
Period: Toddler Dose
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Started | 139 | 139
Vaccination 4 | 139 | 139
Completed | 138 | 138
Not Completed | 1 | 1
Not completed — Withdrawal by parent/guardian | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of study vaccine.
Groups:
- 13vPnC: Multi-dose Vial (With Preservative): Infant series: participants were randomized to receive a single 0.5 mL dose of 13vPnC with preservative 2-PE from a MDV, intramuscularly at age of 6 weeks (Vaccination 1), 10 weeks (Vaccination 2) and 14 weeks (Vaccination 3) along with 2 routine vaccines: 1) DTP-Hib-HBV vaccine, 2) rotavirus vaccine. Participants were followed-up to 1 month after Vaccination 3. Infant series was followed by toddler dose. Toddler dose: participants were administered with a single 0.5 mL dose of 13vPnC vaccine with preservative 2-PE from MDV, intramuscularly at age of 12 months (Vaccination 4) along with routine hepatitis A virus vaccine. Participants were followed-up to 1 month after Vaccination 4. Different limbs were used to administer study vaccine and routine vaccines (according to local clinical practice).
- 13vPnC: Single-dose Prefilled Syringe (Without Preservative): Infant series: participants were randomized to receive a single 0.5 mL dose of 13vPnC without preservative 2-PE from a single-dose PFS, intramuscularly at age of 6 weeks (Vaccination 1), 10 weeks (Vaccination 2) and 14 weeks (Vaccination 3) along with 2 routine vaccines: 1) DTP-Hib-HBV vaccine, 2) rotavirus vaccine. Participants were followed-up to 1 month after Vaccination 3. Infant series was followed by toddler dose. Toddler dose: participants were administered with a single 0.5 mL dose of 13vPnC vaccine without preservative 2-PE from single dose PFS, intramuscularly at age of 12 months (Vaccination 4) along with routine hepatitis A virus vaccine. Participants were followed-up to 1 month after Vaccination 4. Different limbs were used to administer study vaccine and routine vaccines (according to local clinical practice).
- Total: Total of all reporting groups
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative) | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 6.9 (0.95) | 6.9 (0.99) | 6.9 (0.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 67 | 141
  Male | 76 | 83 | 159
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 150 | 150 | 300
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 150 | 150 | 300
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 1
Description: Local reactions were recorded daily using an electronic diary. Local reactions included redness, swelling and pain at injection site. Redness and swelling were graded as mild (0.5 to 2.5 centimeters [cm]), moderate (2.5 to 7.0 cm) and, severe (greater than [>] 7 cm). Pain at injection site was graded as mild (hurt if gently touched (example, whimpers, winces, protests, or withdraws), moderate (hurt if gently touched [with crying]), and severe (caused limitation of limb movement). Participants may be represented in more than 1 row. Here, "Any" for redness, swelling and pain at injection site represents any grade of these local reactions among mild, moderate or severe.
Time Frame: Within 7 days after Vaccination 1
Population: Safety population of infant series included all participants who received at least 1 dose of study vaccine during infant series. Here, "Overall Number of Participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 147 | 148
percentage of participants
  Redness: Any | 19.7 [13.6 to 27.1] | 16.9 [11.2 to 23.9]
  Redness: Mild | 17.7 [11.9 to 24.8] | 12.8 [7.9 to 19.3]
  Redness: Moderate | 2.0 [0.4 to 5.8] | 4.1 [1.5 to 8.6]
  Redness: Severe | 0 [0.0 to 2.5] | 0 [0.0 to 2.5]
  Swelling: Any | 27.9 [20.8 to 35.9] | 33.8 [26.2 to 42.0]
  Swelling: Mild | 21.8 [15.4 to 29.3] | 23.6 [17.1 to 31.3]
  Swelling: Moderate | 6.1 [2.8 to 11.3] | 10.1 [5.8 to 16.2]
  Swelling: Severe | 0 [0.0 to 2.5] | 0 [0.0 to 2.5]
  Pain at injection site: Any | 61.9 [53.5 to 69.8] | 67.6 [59.4 to 75.0]
  Pain at injection site: Mild | 28.6 [21.4 to 36.6] | 33.1 [25.6 to 41.3]
  Pain at injection site: Moderate | 30.6 [23.3 to 38.7] | 29.1 [21.9 to 37.1]
  Pain at injection site: Severe | 2.7 [0.7 to 6.8] | 5.4 [2.4 to 10.4]

2. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 1
Description: Systemic events included fever, decreased appetite, drowsiness(increased sleep) and irritability,were recorded daily using an electronic diary. Fever graded as:1)less than (<)38.0 degrees Celsius [C], 2)greater than or equal to(>=)38.0 degree C to 38.4 degree C, 3)38.5 degree C to 38.9 degree C, 4) 39.0 degree C to 40.0 degree C, 5) >40.0 degree C. Decreased appetite graded as: mild(decreased interest in eating), moderate(decreased oral intake), and severe(refusal to feed). Drowsiness graded as:mild(increased or prolonged sleeping bouts), moderate(slightly subdued; interfering with daily activity), and severe(disabling; not interested in usual daily activity). Irritability graded as: mild(easily consolable), moderate(required increased attention), and severe(inconsolable; crying could not be comforted). Participants may be represented in >1 row. Here,"Any" for decreased appetite, drowsiness, irritability represents any grade of these systemic reactions among mild, moderate or severe.
Time Frame: Within 7 days after Vaccination 1
Population: Safety population for infant series included all participants who received at least 1 dose of study vaccine during infant series. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 147 | 148
percentage of participants
  Fever: <38.0 degree C | 15.0 [9.6 to 21.8] | 10.8 [6.3 to 17.0]
  Fever: >=38.0 degree C to 38.4 degree C | 10.9 [6.4 to 17.1] | 8.1 [4.3 to 13.7]
  Fever: 38.5 degree C to 38.9 degree C | 1.4 [0.2 to 4.8] | 2.7 [0.7 to 6.8]
  Fever: 39.0 degree C to 40.0 degree C | 1.4 [0.2 to 4.8] | 0 [0.0 to 2.5]
  Fever: >40.0 degree C | 1.4 [0.2 to 4.8] | 0 [0.0 to 2.5]
  Decreased appetite: Any | 42.2 [34.1 to 50.6] | 53.4 [45.0 to 61.6]
  Decreased appetite: Mild | 23.8 [17.2 to 31.5] | 30.4 [23.1 to 38.5]
  Decreased appetite: Moderate | 17.7 [11.9 to 24.8] | 21.6 [15.3 to 29.1]
  Decreased appetite: Severe | 0.7 [0.0 to 3.7] | 1.4 [0.2 to 4.8]
  Drowsiness: Any | 55.1 [46.7 to 63.3] | 66.2 [58.0 to 73.8]
  Drowsiness: Mild | 29.3 [22.0 to 37.3] | 33.1 [25.6 to 41.3]
  Drowsiness: Moderate | 25.2 [18.4 to 33.0] | 31.1 [23.7 to 39.2]
  Drowsiness: Severe | 0.7 [0.0 to 3.7] | 2.0 [0.4 to 5.8]
  Irritability: Any | 64.6 [56.3 to 72.3] | 65.5 [57.3 to 73.2]
  Irritability: Mild | 37.4 [29.6 to 45.8] | 32.4 [25.0 to 40.6]
  Irritability: Moderate | 21.8 [15.4 to 29.3] | 26.4 [19.5 to 34.2]
  Irritability: Severe | 5.4 [2.4 to 10.4] | 6.8 [3.3 to 12.1]

3. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 2
Description: Local reactions were recorded daily using an electronic diary. Local reactions included redness, swelling and pain at injection site. Redness and swelling were graded as mild (0.5 to 2.5 cm), moderate (2.5 to 7.0 cm) and, severe (> 7 cm). Pain at injection site was graded as mild (hurt if gently touched (example, whimpers, winces, protests, or withdraws), moderate (hurt if gently touched [with crying]), and severe (caused limitation of limb movement). Participants may be represented in more than 1 row. Here, "Any" for redness, swelling and pain at injection site represents any grade of these local reactions among mild, moderate or severe.
Time Frame: Within 7 days after Vaccination 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 141 | 140
percentage of participants
  Redness: Any | 17.0 [11.2 to 24.3] | 19.3 [13.1 to 26.8]
  Redness: Mild | 16.3 [10.6 to 23.5] | 17.9 [11.9 to 25.2]
  Redness: Moderate | 0.7 [0.0 to 3.9] | 1.4 [0.2 to 5.1]
  Redness: Severe | 0 [0.0 to 2.6] | 0 [0.0 to 2.6]
  Swelling: Any | 24.8 [17.9 to 32.8] | 27.9 [20.6 to 36.1]
  Swelling: Mild | 21.3 [14.8 to 29.0] | 22.9 [16.2 to 30.7]
  Swelling: Moderate | 3.5 [1.2 to 8.1] | 5.0 [2.0 to 10.0]
  Swelling: Severe | 0 [0.0 to 2.6] | 0 [0.0 to 2.6]
  Pain at injection site: Any | 59.6 [51.0 to 67.7] | 62.1 [53.6 to 70.2]
  Pain at injection site: Mild | 32.6 [25.0 to 41.0] | 29.3 [21.9 to 37.6]
  Pain at injection site: Moderate | 20.6 [14.2 to 28.2] | 26.4 [19.3 to 34.5]
  Pain at injection site: Severe | 6.4 [3.0 to 11.8] | 6.4 [3.0 to 11.9]

4. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 2
Description: Systemic events included fever, decreased appetite, drowsiness(increased sleep) and irritability, were recorded daily using an electronic diary. Fever graded as:1) < 38.0 degrees C, 2) >= 38.0 degree C to 38.4 degree C, 3)38.5 degree C to 38.9 degree C, 4) 39.0 degree C to 40.0 degree C, 5) >40.0 degree C. Decreased appetite graded as: mild(decreased interest in eating), moderate(decreased oral intake), and severe(refusal to feed). Drowsiness graded as: mild (increased or prolonged sleeping bouts), moderate (slightly subdued; interfering with daily activity), and severe (disabling; not interested in usual daily activity). Irritability graded as: mild (easily consolable), moderate (required increased attention), and severe (inconsolable; crying could not be comforted). Participants may be represented in >1 row. Here, "Any" for decreased appetite, drowsiness, irritability represents any grade of these systemic reactions among mild, moderate or severe.
Time Frame: Within 7 days after Vaccination 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 141 | 140
percentage of participants
  Fever: <38.0 degree C | 8.5 [4.5 to 14.4] | 8.6 [4.5 to 14.5]
  Fever: >=38.0 degree C to 38.4 degree C | 6.4 [3.0 to 11.8] | 5.7 [2.5 to 10.9]
  Fever: 38.5 degree C to 38.9 degree C | 2.1 [0.4 to 6.1] | 2.1 [0.4 to 6.1]
  Fever: 39.0 degree C to 40.0 degree C | 0 [0.0 to 2.6] | 0 [0.0 to 2.6]
  Fever: >40.0 degree C | 0 [0.0 to 2.6] | 0.7 [0.0 to 3.9]
  Decreased appetite: Any | 40.4 [32.3 to 49.0] | 38.6 [30.5 to 47.2]
  Decreased appetite: Mild | 27.0 [19.8 to 35.1] | 25.0 [18.1 to 33.0]
  Decreased appetite: Moderate | 12.1 [7.2 to 18.6] | 12.1 [7.2 to 18.7]
  Decreased appetite: Severe | 1.4 [0.2 to 5.0] | 1.4 [0.2 to 5.1]
  Drowsiness: Any | 50.4 [41.8 to 58.9] | 52.1 [43.5 to 60.7]
  Drowsiness: Mild | 23.4 [16.7 to 31.3] | 22.1 [15.6 to 29.9]
  Drowsiness: Moderate | 25.5 [18.6 to 33.6] | 26.4 [19.3 to 34.5]
  Drowsiness: Severe | 1.4 [0.2 to 5.0] | 3.6 [1.2 to 8.1]
  Irritability: Any | 56.7 [48.1 to 65.0] | 60.0 [51.4 to 68.2]
  Irritability: Mild | 29.1 [21.7 to 37.3] | 37.9 [29.8 to 46.4]
  Irritability: Moderate | 24.8 [17.9 to 32.8] | 17.9 [11.9 to 25.2]
  Irritability: Severe | 2.8 [0.8 to 7.1] | 4.3 [1.6 to 9.1]

5. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 3
Description: as for outcome 3
Time Frame: Within 7 days after Vaccination 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 139 | 140
percentage of participants
  Redness: Any | 20.1 [13.8 to 27.8] | 22.9 [16.2 to 30.7]
  Redness: Mild | 20.1 [13.8 to 27.8] | 20.0 [13.7 to 27.6]
  Redness: Moderate | 0 [0.0 to 2.6] | 2.9 [0.8 to 7.2]
  Redness: Severe | 0 [0.0 to 2.6] | 0 [0.0 to 2.6]
  Swelling: Any | 23.0 [16.3 to 30.9] | 27.1 [20.0 to 35.3]
  Swelling: Mild | 20.9 [14.4 to 28.6] | 23.6 [16.8 to 31.5]
  Swelling: Moderate | 2.2 [0.4 to 6.2] | 2.9 [0.8 to 7.2]
  Swelling: Severe | 0 [0.0 to 2.6] | 0.7 [0.0 to 3.9]
  Pain at injection site: Any | 55.4 [46.7 to 63.8] | 54.3 [45.7 to 62.7]
  Pain at injection site: Mild | 30.2 [22.7 to 38.6] | 27.9 [20.6 to 36.1]
  Pain at injection site: Moderate | 23.0 [16.3 to 30.9] | 21.4 [14.9 to 29.2]
  Pain at injection site: Severe | 2.2 [0.4 to 6.2] | 5.0 [2.0 to 10.0]

6. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 3
Description: as for outcome 4
Time Frame: Within 7 days after Vaccination 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 139 | 140
percentage of participants
  Fever: <38.0 degree C | 7.2 [3.5 to 12.8] | 9.3 [5.0 to 15.4]
  Fever: >=38.0 degree C to 38.4 degree C | 4.3 [1.6 to 9.2] | 6.4 [3.0 to 11.9]
  Fever: 38.5 degree C to 38.9 degree C | 2.2 [0.4 to 6.2] | 1.4 [0.2 to 5.1]
  Fever: 39.0 degree C to 40.0 degree C | 0 [0.0 to 2.6] | 1.4 [0.2 to 5.1]
  Fever: >40.0 degree C | 0.7 [0.0 to 3.9] | 0 [0.0 to 2.6]
  Decreased appetite: Any | 34.5 [26.7 to 43.1] | 36.4 [28.5 to 45.0]
  Decreased appetite: Mild | 20.1 [13.8 to 27.8] | 23.6 [16.8 to 31.5]
  Decreased appetite: Moderate | 11.5 [6.7 to 18.0] | 10.0 [5.6 to 16.2]
  Decreased appetite: Severe | 2.9 [0.8 to 7.2] | 2.9 [0.8 to 7.2]
  Drowsiness: Any | 36.0 [28.0 to 44.5] | 39.3 [31.1 to 47.9]
  Drowsiness: Mild | 20.9 [14.4 to 28.6] | 19.3 [13.1 to 26.8]
  Drowsiness: Moderate | 13.7 [8.4 to 20.5] | 17.9 [11.9 to 25.2]
  Drowsiness: Severe | 1.4 [0.2 to 5.1] | 2.1 [0.4 to 6.1]
  Irritability: Any | 54.7 [46.0 to 63.1] | 60.0 [51.4 to 68.2]
  Irritability: Mild | 31.7 [24.0 to 40.1] | 37.9 [29.8 to 46.4]
  Irritability: Moderate | 19.4 [13.2 to 27.0] | 15.7 [10.1 to 22.8]
  Irritability: Severe | 3.6 [1.2 to 8.2] | 6.4 [3.0 to 11.9]

7. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 4
Description: as for outcome 3
Time Frame: Within 7 days after Vaccination 4
Population: Safety population for toddler dose included all participants who received at least 1 dose of study vaccine during toddler dosing. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 132 | 132
percentage of participants
  Redness: Any | 8.3 [4.2 to 14.4] | 11.4 [6.5 to 18.0]
  Redness: MIld | 8.3 [4.2 to 14.4] | 10.6 [5.9 to 17.2]
  Redness: Moderate | 0 [0.0 to 2.8] | 0.8 [0.0 to 4.1]
  Redness: Severe | 0 [0.0 to 2.8] | 0 [0.0 to 2.8]
  Swelling: Any | 9.1 [4.8 to 15.3] | 12.1 [7.1 to 18.9]
  Swelling: Mild | 6.8 [3.2 to 12.5] | 11.4 [6.5 to 18.0]
  Swelling: Moderate | 2.3 [0.5 to 6.5] | 0.8 [0.0 to 4.1]
  Swelling: Severe | 0 [0.0 to 2.8] | 0 [0.0 to 2.8]
  Pain at injection site: Any | 25.0 [17.9 to 33.3] | 19.7 [13.3 to 27.5]
  Pain at injection site: Mild | 18.9 [12.6 to 26.7] | 13.6 [8.3 to 20.7]
  Pain at injection site: Moderate | 6.1 [2.7 to 11.6] | 5.3 [2.2 to 10.6]
  Pain at injection site: Severe | 0 [0.0 to 2.8] | 0.8 [0.0 to 4.1]

8. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 4
Description: as for outcome 4
Time Frame: Within 7 days after Vaccination 4
Population: Safety population for toddler dose included all participants who received at least 1 dose of study vaccine during toddler dosing. Here, "Overall Number of Participants Analyzed, N" signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 132 | 132
percentage of participants
  Fever: <38.0 degree C | 3.0 [0.8 to 7.6] | 4.5 [1.7 to 9.6]
  Fever: >=38.0 degree C to 38.4 degree C | 1.5 [0.2 to 5.4] | 3.8 [1.2 to 8.6]
  Fever: 38.5 degree C to 38.9 degree C | 0 [0.0 to 2.8] | 0 [0.0 to 2.8]
  Fever: 39.0 degree C to 40.0 degree C | 0 [0.0 to 2.8] | 0.8 [0.0 to 4.1]
  Fever: >40.0 degree C | 1.5 [0.2 to 5.4] | 0 [0.0 to 2.8]
  Decreased appetite: Any | 15.2 [9.5 to 22.4] | 16.7 [10.7 to 24.1]
  Decreased appetite: Mild | 10.6 [5.9 to 17.2] | 6.8 [3.2 to 12.5]
  Decreased appetite: Moderate | 4.5 [1.7 to 9.6] | 9.8 [5.3 to 16.3]
  Decreased appetite: Severe | 0 [0.0 to 2.8] | 0 [0.0 to 2.8]
  Drowsiness: Any | 7.6 [3.7 to 13.5] | 18.9 [12.6 to 26.7]
  Drowsiness: Mild | 3.8 [1.2 to 8.6] | 12.9 [7.7 to 19.8]
  Drowsiness: Moderate | 3.8 [1.2 to 8.6] | 6.1 [2.7 to 11.6]
  Drowsiness: Severe | 0 [0.0 to 2.8] | 0 [0.0 to 2.8]
  Irritability: Any | 24.2 [17.2 to 32.5] | 23.5 [16.5 to 31.6]
  Irritability: Mild | 15.9 [10.1 to 23.3] | 16.7 [10.7 to 24.1]
  Irritability: Moderate | 7.6 [3.7 to 13.5] | 5.3 [2.2 to 10.6]
  Irritability: Severe | 0.8 [0.0 to 4.1] | 1.5 [0.2 to 5.4]

9. Primary Outcome: Percentage of Participants With Adverse Events (AEs) After Vaccination 1 up to 1 Month After Vaccination 3
Description: An AE was any untoward medical occurrence in a participant who received study vaccine without regard to possibility of causal relationship.
Time Frame: From Vaccination 1 up to 1 Month after Vaccination 3 (for a maximum study duration of 3 months)
Population: Safety population for infant series included all participants who received at least 1 dose of study vaccine during infant series.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 150 | 150
percentage of participants | 47.3 [39.1 to 55.6] | 49.3 [41.1 to 57.6]

10. Primary Outcome: Percentage of Participants With Adverse Events (AEs) From Vaccination 4 up to 1 Month After Vaccination 4
Description: as for outcome 9
Time Frame: From Vaccination 4 up to 1 month after Vaccination 4 (for a maximum study duration of 1 month)
Population: Safety population for toddler dose included all participants who received at least 1 dose of study vaccine during toddler dosing.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 139 | 139
percentage of participants | 7.9 [4.0 to 13.7] | 8.6 [4.5 to 14.6]

11. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) After Vaccination 1 up to 1 Month After Vaccination 4
Description: An AE was any untoward medical occurrence in a participant who received study vaccine without regard to possibility of causal relationship. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: From Vaccination 1 up to 1 month after Vaccination 4 (for a maximum study duration of 11.5 months)
Population: Safety population included all participants who received at least 1 dose of study vaccine in study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 13vPnC: Multi-dose Vial (With Preservative): This arm represents the combined Infant series and Toddler dose. Infant series: participants were randomized to receive a single 0.5 mL dose of 13vPnC with preservative 2-PE from a MDV, intramuscularly at age of 6 weeks (Vaccination 1), 10 weeks (Vaccination 2) and 14 weeks (Vaccination 3) along with 2 routine vaccines: 1) DTP-Hib-HBV vaccine, 2) rotavirus vaccine. Participants were followed-up to 1 month after Vaccination 3. Infant series was followed by toddler dose. Toddler dose: participants were administered with a single 0.5 mL dose of 13vPnC vaccine with preservative 2-PE from MDV, intramuscularly at age of 12 months (Vaccination 4) along with routine hepatitis A virus vaccine. Participants were followed-up to 1 month after Vaccination 4. Different limbs were used to administer study vaccine and routine vaccines (according to local clinical practice).
- 13vPnC: Single-dose Prefilled Syringe (Without Preservative): This arm represents the combined Infant series and Toddler dose. Infant series: participants were randomized to receive a single 0.5 mL dose of 13vPnC without preservative 2-PE from a single-dose PFS, intramuscularly at age of 6 weeks (Vaccination 1), 10 weeks (Vaccination 2) and 14 weeks (Vaccination 3) along with 2 routine vaccines: 1) DTP-Hib-HBV vaccine, 2) rotavirus vaccine. Participants were followed-up to 1 month after Vaccination 3. Infant series was followed by toddler dose. Toddler dose: participants were administered with a single 0.5 mL dose of 13vPnC vaccine without preservative 2-PE from single dose PFS, intramuscularly at age of 12 months (Vaccination 4) along with routine hepatitis A virus vaccine. Participants were followed-up to 1 month after Vaccination 4. Different limbs were used to administer study vaccine and routine vaccines (according to local clinical practice).
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 150 | 150
percentage of participants | 8.0 [4.2 to 13.6] | 4.7 [1.9 to 9.4]

12. Primary Outcome: Number of Participants With New Diagnosed Chronic Medical Condition (NDCMC) From 1 Month After Vaccination 3 up to Vaccination 4
Description: A newly diagnosed chronic medical condition was defined as a disease or medical condition, not previously identified, that was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: From 1 month after Vaccination 3 up to Vaccination 4 (for a maximum study duration of 7.5 months)
Population: Safety population for study included all participants who received at least 1 dose of study vaccine in study.
Measure: Count of Participants; unit: Participants
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 150 | 150
Participants | 0 | 0

13. Secondary Outcome: Percentage of Participants With Immunoglobulin G (IgG) Concentrations Greater Than or Equal to (>=) Pre-defined Thresholds for Each of the Pneumococcal Serotypes Measured 1 Month After Vaccination 3
Description: Percentage of participants achieving predefined antibody threshold: >=0.35 microgram per milliliter (mcg/mL) for the 10 pneumococcal serotypes 1, 3, 4, 6A, 7F, 9V, 14, 18C, 19F and 23F; threshold >= 0.23 mcg/mL for serotype 5, threshold >= 0.10 mcg/mL for serotype 6B, threshold >= 0.12 mcg/mL for serotype 19A, along with the corresponding 95 percent (%) confidence interval (CI) are reported.
Time Frame: 1 month after Vaccination 3
Population: Evaluable immunogenicity population(EIP) for infant series: all eligible participants aged 6 weeks at time of Dose 1, who received 3 doses of infant series vaccine, had blood drawn post Dose 3 within 27 to 56 days(inclusive) post Dose 3, had at least 1 valid and determinate assay result post Dose 3, and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 136 | 133
percentage of participants
  Serotype: 1 | 91.2 [85.1 to 95.4] | 85.0 [77.7 to 90.6]
  Serotype: 3 | 91.9 [86.0 to 95.9] | 85.7 [78.6 to 91.2]
  Serotype: 4 | 91.2 [85.1 to 95.4] | 91.0 [84.8 to 95.3]
  Serotype: 5 | 84.6 [77.4 to 90.2] | 82.0 [74.4 to 88.1]
  Serotype: 6A | 83.8 [76.5 to 89.6] | 71.4 [63.0 to 78.9]
  Serotype: 6B | 77.2 [69.2 to 84.0] | 75.2 [67.0 to 82.3]
  Serotype: 7F | 96.3 [91.6 to 98.8] | 93.2 [87.5 to 96.9]
  Serotype: 9V | 85.3 [78.2 to 90.8] | 83.5 [76.0 to 89.3]
  Serotype: 14 | 88.2 [81.6 to 93.1] | 82.7 [75.2 to 88.7]
  Serotype: 18C | 92.6 [86.9 to 96.4] | 84.2 [76.9 to 90.0]
  Serotype: 19A | 100.0 [97.3 to 100.0] | 98.5 [94.7 to 99.8]
  Serotype: 19F | 97.8 [93.7 to 99.5] | 95.5 [90.4 to 98.3]
  Serotype: 23F | 84.6 [77.4 to 90.2] | 76.7 [68.6 to 83.6]

14. Secondary Outcome: Percentage of Participants With Immunoglobulin G (IgG) Concentrations Greater Than or Equal to (>=) Pre-defined Thresholds for Each of the Pneumococcal Serotypes Measured 1 Month After Vaccination 4
Description: Percentage of participants achieving predefined antibody threshold >=0.35 mcg/mL for the 10 pneumococcal serotypes 1, 3, 4, 6A, 7F, 9V, 14, 18C, 19F and 23F, threshold >= 0.23 mcg/mL for serotype 5, threshold >= 0.10 mcg/mL for serotype 6B, threshold >= 0.12 mcg/mL for serotype 19A, along with the corresponding 95% CI are reported.
Time Frame: 1 month after Vaccination 4
Population: EIP for toddler dose: all eligible participants who received 3 doses in infant series and 1 toddler dose of vaccine, had blood drawn post Dose 4 within 27 to 56 days (inclusive) post Dose 4, had at least 1 valid and determinate assay result post Dose 4, and had no major protocol violations. "N": signifies participants evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 132 | 129
percentage of participants
  Serotype: 1 | 99.2 [95.9 to 100.0] | 100.0 [97.2 to 100.0]
  Serotype: 3 | 97.0 [92.4 to 99.2] | 98.4 [94.5 to 99.8]
  Serotype: 4 | 99.2 [95.9 to 100.0] | 100.0 [97.2 to 100.0]
  Serotype: 5 | 99.2 [95.9 to 100.0] | 100.0 [97.2 to 100.0]
  Serotype: 6A | 96.2 [91.4 to 98.8] | 96.9 [92.3 to 99.1]
  Serotype: 6B | 98.5 [94.6 to 99.8] | 96.9 [92.3 to 99.1]
  Serotype: 7F | 99.2 [95.9 to 100.0] | 99.2 [95.8 to 100.0]
  Serotype: 9V | 98.5 [94.6 to 99.8] | 99.2 [95.8 to 100.0]
  Serotype: 14 | 97.7 [93.5 to 99.5] | 96.1 [91.2 to 98.7]
  Serotype: 18C | 97.0 [92.4 to 99.2] | 99.2 [95.8 to 100.0]
  Serotype: 19A | 99.2 [95.9 to 100.0] | 99.2 [95.8 to 100.0]
  Serotype: 19F | 98.5 [94.6 to 99.8] | 100.0 [97.2 to 100.0]
  Serotype: 23F | 99.2 [95.9 to 100.0] | 96.9 [92.3 to 99.1]

15. Secondary Outcome: Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) for Each of Pneumococcal Serotypes Measured 1 Month After Vaccination 3
Description: Antibody (IgG) GMCs for the 13 pneumococcal serotypes (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F) and corresponding 2-sided 95% CI are reported.
Time Frame: 1 month after Vaccination 3
Population: Evaluable immunogenicity population for infant series: all eligible participants aged 6 weeks at time of Dose 1, who received 3 doses of infant series vaccine, had blood drawn post-Dose 3 within 27 to 56 days (inclusive) post Dose 3, had at least 1 valid and determinate assay result post Dose 3, and had no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 136 | 133
mcg/mL
  Serotype: 1 | 1.36 [1.15 to 1.60] | 1.13 [0.94 to 1.36]
  Serotype: 3 | 1.01 [0.88 to 1.16] | 0.93 [0.80 to 1.07]
  Serotype: 4 | 1.67 [1.40 to 1.98] | 1.75 [1.45 to 2.11]
  Serotype: 5 | 0.83 [0.67 to 1.02] | 0.86 [0.67 to 1.11]
  Serotype: 6A | 1.45 [1.13 to 1.87] | 0.86 [0.66 to 1.12]
  Serotype: 6B | 0.41 [0.31 to 0.55] | 0.33 [0.24 to 0.46]
  Serotype: 7F | 2.01 [1.74 to 2.33] | 1.85 [1.52 to 2.26]
  Serotype: 9V | 1.42 [1.17 to 1.73] | 1.28 [1.02 to 1.62]
  Serotype: 14 | 1.66 [1.33 to 2.06] | 1.39 [1.09 to 1.76]
  Serotype: 18C | 1.81 [1.50 to 2.18] | 1.37 [1.10 to 1.71]
  Serotype: 19A | 2.33 [1.96 to 2.78] | 1.86 [1.51 to 2.28]
  Serotype: 19F | 2.89 [2.52 to 3.31] | 2.43 [2.04 to 2.89]
  Serotype: 23F | 1.48 [1.20 to 1.81] | 0.94 [0.73 to 1.21]

16. Secondary Outcome: Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) for Each of Pneumococcal Serotypes Measured 1 Month After Vaccination 4
Description: as for outcome 15
Time Frame: 1 month after Vaccination 4
Population: Evaluable immunogenicity population for toddler dose: all eligible participants who received 3 doses in infant series and 1 toddler dose of vaccine, had blood drawn post Dose 4 within 27 to 56 days (inclusive) post Dose 4, had at least 1 valid and determinate assay result post Dose 4, and had no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 132 | 130
mcg/mL
  Serotype: 1 | 4.35 [3.71 to 5.10] | 4.27 [3.65 to 4.99]
  Serotype: 3 | 1.58 [1.36 to 1.83] | 1.63 [1.43 to 1.86]
  Serotype: 4 | 10.58 [8.89 to 12.60] | 11.91 [10.19 to 13.93]
  Serotype: 5 | 5.16 [4.37 to 6.10] | 5.68 [4.81 to 6.70]
  Serotype: 6A | 18.55 [14.32 to 24.02] | 20.51 [16.32 to 25.78]
  Serotype: 6B | 11.76 [9.24 to 14.98] | 10.87 [8.14 to 14.53]
  Serotype: 7F | 7.92 [6.88 to 9.13] | 8.29 [7.17 to 9.57]
  Serotype: 9V | 8.78 [7.19 to 10.73] | 9.57 [8.00 to 11.44]
  Serotype: 14 | 13.20 [10.69 to 16.30] | 11.78 [9.31 to 14.90]
  Serotype: 18C | 6.21 [5.19 to 7.44] | 6.27 [5.25 to 7.48]
  Serotype: 19A | 12.26 [10.26 to 14.65] | 12.02 [9.75 to 14.82]
  Serotype: 19F | 13.65 [11.16 to 16.69] | 14.09 [11.71 to 16.96]
  Serotype: 23F | 10.89 [8.78 to 13.50] | 9.90 [7.75 to 12.66]

17. Secondary Outcome: Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) for Each of Pneumococcal Serotypes Measured 1 Month After Vaccination 3
Description: Antibody-mediated serum OPA against the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) was measured centrally using a pneumococcal OPA assay. Initial results were measured as OPA titers, which were then logarithmically transformed for analysis; geometric means calculated and expressed as GMTs.
Time Frame: 1 month after Vaccination 3
Population: Evaluable immunogenicity population for infant series: all eligible participants aged 6 weeks at time of Dose 1, who received 3 doses of infant series vaccine, had blood drawn post Dose 3 within 27 to 56 days (inclusive) post Dose 3, had at least 1 valid and determinate assay result post Dose 3, and had no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: titer (1/dilution)
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 136 | 133
titer (1/dilution)
  Serotype: 1 | 21.8 [18.1 to 26.2] | 22.5 [18.1 to 27.9]
  Serotype: 3 | 79.7 [68.8 to 92.3] | 72.8 [62.7 to 84.6]
  Serotype: 4 | 1158.8 [938.3 to 1431.1] | 1159.2 [948.3 to 1417.0]
  Serotype: 5 | 37.0 [31.4 to 43.5] | 40.9 [34.0 to 49.3]
  Serotype: 6A | 1211.7 [896.4 to 1638.0] | 1321.9 [1026.7 to 1701.9]
  Serotype: 6B | 1145.8 [870.4 to 1508.3] | 957.6 [708.2 to 1294.8]
  Serotype: 7F | 1743.3 [1436.6 to 2115.5] | 1178.8 [952.6 to 1458.6]
  Serotype: 9V | 643.9 [498.6 to 831.7] | 683.3 [522.6 to 893.3]
  Serotype: 14 | 496.9 [344.2 to 717.3] | 341.8 [236.0 to 495.0]
  Serotype: 18C | 3055.8 [2378.5 to 3926.0] | 2183.9 [1686.9 to 2827.3]
  Serotype: 19A | 219.3 [169.4 to 283.9] | 275.7 [212.0 to 358.6]
  Serotype: 19F | 236.1 [191.6 to 291.1] | 272.7 [219.1 to 339.4]
  Serotype: 23F | 1036.4 [746.9 to 1438.0] | 926.8 [673.9 to 1274.7]

18. Secondary Outcome: Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMT) for Each of Pneumococcal Serotypes Measured 1 Month After Vaccination 4
Description: as for outcome 17
Time Frame: 1 month after Vaccination 4
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: titer (1/dilution)
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 132 | 130
titer (1/dilution)
  Serotype: 1 | 204.2 [164.7 to 253.3] | 217.0 [176.4 to 266.9]
  Serotype: 3 | 121.0 [104.4 to 140.3] | 129.8 [111.7 to 150.8]
  Serotype: 4 | 2991.4 [2437.5 to 3671.3] | 2519.0 [2098.7 to 3023.6]
  Serotype: 5 | 157.6 [131.9 to 188.3] | 153.4 [126.6 to 185.8]
  Serotype: 6A | 2945.7 [2376.0 to 3652.1] | 3092.5 [2493.5 to 3835.4]
  Serotype: 6B | 1948.9 [1521.4 to 2496.7] | 1750.1 [1360.9 to 2250.8]
  Serotype: 7F | 4161.5 [3498.0 to 4950.9] | 4353.8 [3706.5 to 5114.0]
  Serotype: 9V | 6927.5 [5765.9 to 8323.2] | 6460.4 [5277.3 to 7908.7]
  Serotype: 14 | 1505.8 [1246.5 to 1819.0] | 1302.2 [1106.1 to 1533.2]
  Serotype: 18C | 8028.3 [6233.7 to 10339.7] | 7830.0 [5998.5 to 10220.7]
  Serotype: 19A | 1848.9 [1472.0 to 2322.2] | 1832.5 [1454.9 to 2308.1]
  Serotype: 19F | 808.0 [633.0 to 1033.5] | 766.0 [609.2 to 963.2]
  Serotype: 23F | 3125.0 [2450.8 to 3984.7] | 3348.8 [2639.5 to 4248.5]

19. Secondary Outcome: Percentage of Participants With Opsonophagocytic Activity (OPA) Titers >= Lower Limit of Quantitation (LLOQ) for Each of Pneumococcal Serotypes Measured 1 Month After Vaccination 3
Description: Percentage of participants achieving OPA titer >=LLOQ along with 95% CI for the 13 pneumococcal serotypes (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F) determined in blood samples of participants was presented. LLOQ (measured in mcg/mL) for each serotype is as follows: Serotype 1=18; Serotype 3=12; Serotype 4=21; Serotype 5=29; Serotype 6A=37; Serotype 6B=43; Serotype 7F=113; Serotype 9V=141; Serotype 14=35; Serotype 18C=31; Serotype 19A=18; Serotype 19F=48; Serotype 23F=13.
Time Frame: 1 month after Vaccination 3
Population: Evaluable immunogenicity population for infant series was analyzed. "Overall Number of Participants Analyzed": signifies participants evaluable for this outcome measure. "Number Analyzed": signifies participants evaluable for specific serotype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 114 | 108
percentage of participants
  Serotype: 1: number analyzed (Participants) | 111 | 106
  Serotype: 1 | 51.4 [41.7 to 61.0] | 46.2 [36.5 to 56.2]
  Serotype: 3: number analyzed (Participants) | 109 | 107
  Serotype: 3 | 98.2 [93.5 to 99.8] | 98.1 [93.4 to 99.8]
  Serotype: 4: number analyzed (Participants) | 105 | 101
  Serotype: 4 | 98.1 [93.3 to 99.8] | 99.0 [94.6 to 100.0]
  Serotype: 5: number analyzed (Participants) | 114 | 107
  Serotype: 5 | 62.3 [52.7 to 71.2] | 62.6 [52.7 to 71.8]
  Serotype: 6A: number analyzed (Participants) | 113 | 107
  Serotype: 6A | 91.2 [84.3 to 95.7] | 94.4 [88.2 to 97.9]
  Serotype: 6B: number analyzed (Participants) | 109 | 104
  Serotype: 6B | 94.5 [88.4 to 98.0] | 92.3 [85.4 to 96.6]
  Serotype: 7F: number analyzed (Participants) | 96 | 93
  Serotype: 7F | 99.0 [94.3 to 100.0] | 96.8 [90.9 to 99.3]
  Serotype: 9V: number analyzed (Participants) | 103 | 100
  Serotype: 9V | 88.3 [80.5 to 93.8] | 88.0 [80.0 to 93.6]
  Serotype: 14: number analyzed (Participants) | 111 | 108
  Serotype: 14 | 82.9 [74.6 to 89.4] | 76.9 [67.8 to 84.4]
  Serotype: 18C: number analyzed (Participants) | 103 | 99
  Serotype: 18C | 98.1 [93.2 to 99.8] | 98.0 [92.9 to 99.8]
  Serotype: 19A: number analyzed (Participants) | 101 | 92
  Serotype: 19A | 92.1 [85.0 to 96.5] | 95.7 [89.2 to 98.8]
  Serotype: 19F: number analyzed (Participants) | 107 | 105
  Serotype: 19F | 89.7 [82.3 to 94.8] | 91.4 [84.4 to 96.0]
  Serotype: 23F: number analyzed (Participants) | 99 | 98
  Serotype: 23F | 94.9 [88.6 to 98.3] | 94.9 [88.5 to 98.3]

20. Secondary Outcome: Percentage of Participants With Opsonophagocytic Activity (OPA) Titers >= Lower Limit of Quantitation (LLOQ) for Each of Pneumococcal Serotypes Measured 1 Month After Vaccination 4
Description: as for outcome 19
Time Frame: 1 month after Vaccination 4
Population: Evaluable immunogenicity population for toddler dose was analyzed. "Overall Number of Participants Analyzed": signifies participants evaluable for this outcome measure. "Number Analyzed": signifies participants evaluable for specific serotype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC: Multi-dose Vial (With Preservative) | 13vPnC: Single-dose Prefilled Syringe (Without Preservative)
Number analyzed (Participants) | 106 | 102
percentage of participants
  Serotype: 1: number analyzed (Participants) | 105 | 102
  Serotype: 1 | 97.1 [91.9 to 99.4] | 97.1 [91.6 to 99.4]
  Serotype: 3: number analyzed (Participants) | 106 | 101
  Serotype: 3 | 98.1 [93.4 to 99.8] | 100.0 [96.4 to 100.0]
  Serotype: 4: number analyzed (Participants) | 102 | 99
  Serotype: 4 | 100.0 [96.4 to 100.0] | 100.0 [96.3 to 100.0]
  Serotype: 5: number analyzed (Participants) | 105 | 102
  Serotype: 5 | 95.2 [89.2 to 98.4] | 97.1 [91.6 to 99.4]
  Serotype: 6A: number analyzed (Participants) | 104 | 101
  Serotype: 6A | 100.0 [96.5 to 100.0] | 99.0 [94.6 to 100.0]
  Serotype: 6B: number analyzed (Participants) | 101 | 101
  Serotype: 6B | 97.0 [91.6 to 99.4] | 95.0 [88.8 to 98.4]
  Serotype: 7F: number analyzed (Participants) | 97 | 90
  Serotype: 7F | 100.0 [96.3 to 100.0] | 100.0 [96.0 to 100.0]
  Serotype: 9V: number analyzed (Participants) | 100 | 98
  Serotype: 9V | 100.0 [96.4 to 100.0] | 99.0 [94.4 to 100.0]
  Serotype: 14: number analyzed (Participants) | 106 | 101
  Serotype: 14 | 100.0 [96.6 to 100.0] | 100.0 [96.4 to 100.0]
  Serotype: 18C: number analyzed (Participants) | 100 | 100
  Serotype: 18C | 99.0 [94.6 to 100.0] | 99.0 [94.6 to 100.0]
  Serotype: 19A: number analyzed (Participants) | 97 | 96
  Serotype: 19A | 100.0 [96.3 to 100.0] | 99.0 [94.3 to 100.0]
  Serotype: 19F: number analyzed (Participants) | 102 | 99
  Serotype: 19F | 96.1 [90.3 to 98.9] | 97.0 [91.4 to 99.4]
  Serotype: 23F: number analyzed (Participants) | 102 | 96
  Serotype: 23F | 99.0 [94.7 to 100.0] | 99.0 [94.3 to 100.0]

ADVERSE EVENTS:
Time Frame: Infant series: SAEs and non-SAEs= from Vaccination 1 up to 1 month post Vaccination 3 (for 3 months). Between infant series and toddler dose: SAEs:1 month post Vaccination 3 up to pre-vaccination 4 (for 7.5 months), non-SAEs were not planned to be collected. Toddler dose: SAEs and non-SAEs = up to 1 month post Vaccination 4 (for 1 month). Local reactions and systemic events =7 days post any vaccination (systematic assessment)
Description: AE term can be both SAE and non-SAE, but are distinct events. Participant may have an event both as SAE and non-SAE. Safety population evaluated. Participants in infant series were followed up from Vaccination 1 till pre-vaccination 4 (toddler dose) irrespective of dose received in infant series, so counted in arms: "13vPnC, MDV: Between Infant Series And Toddler Dose" and "13vPnC, PFS: Between Infant Series and Toddler Dose". Toddler dose series included 139 participants who had Vaccination 4.
Groups:
- 13vPnC, MDV With Preservative: Infant Series: Infant series: participants were randomized to receive a single 0.5 mL dose of 13vPnC with preservative 2-PE from a MDV, intramuscularly at age of 6 weeks (Vaccination 1), 10 weeks (Vaccination 2) and 14 weeks (Vaccination 3) respectively along with 2 routine vaccines: 1) DTP-Hib-HBV vaccine, 2) rotavirus vaccine. Participants were followed-up to 1 month after Vaccination 3. Different limbs were used to administer study vaccine and routine vaccines (according to local clinical practice).
- 13vPnC, PFS Without Preservative: Infant Series: Infant series: participants were randomized to receive a single 0.5 mL dose of 13vPnC without preservative 2-PE from a single dose PFS, intramuscularly at age of 6 weeks (Vaccination 1), 10 weeks (Vaccination 2) and 14 weeks (Vaccination 3) respectively along with 2 routine vaccines: 1) DTP-Hib-HBV vaccine, 2) rotavirus vaccine. Participants were followed-up to 1 month after Vaccination 3. Different limbs were used to administer study vaccine and routine vaccines (according to local clinical practice).
- 13vPnC, MDV: Between Infant Series and Toddler Dose: This arm is created to report the safety data of participants for the duration "from 1 month after infant series until the time of toddler dose vaccination (pre-vaccination)". It included participants who received any dose of 13vPnC vaccine with preservative 2-PE from a MDV, intramuscularly during infant series and followed up to vaccination in toddler dose.
- 13vPnC, PFS: Between Infant Series and Toddler Dose: This arm is created to report the safety data of participants for the duration "from 1 month after infant series until the time of toddler dose vaccination (pre-vaccination)". It included participants who received any dose of 13vPnC vaccine without preservative 2-PE from a single dose PFS, intramuscularly during infant series and followed up to vaccination in toddler dose.
- 13vPnC, MDV With Preservative: Toddler Dose: Toddler dose followed infant series. Toddler dose: participants were administered a single 0.5 mL dose of 13vPnC vaccine with preservative 2-PE from a MDV intramuscularly, at age of 12 months (Vaccination 4) along with routine hepatitis A virus vaccine. Participants were followed-up to 1 month after Vaccination 4. Different limbs were used to administer study vaccine and routine vaccines (according to local clinical practice).
- 13vPnC, PFS Without Preservative: Toddler Dose: Toddler dose followed infant series. Toddler dose: participants were administered a single 0.5 mL dose of 13vPnC vaccine without preservative 2-PE from a single- dose PFS, at age of 12 months (Vaccination 4) along with routine hepatitis A virus vaccine. Participants were followed-up to 1 month after Vaccination 4. Different limbs were used to administer study vaccine and routine vaccines (according to local clinical practice).
Arm/Group | 13vPnC, MDV With Preservative: Infant Series | 13vPnC, PFS Without Preservative: Infant Series | 13vPnC, MDV: Between Infant Series and Toddler Dose | 13vPnC, PFS: Between Infant Series and Toddler Dose | 13vPnC, MDV With Preservative: Toddler Dose | 13vPnC, PFS Without Preservative: Toddler Dose
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/150 | 0/150 | 0/150 | 0/139 | 0/139
Serious Adverse Events (participants affected / at risk) | 5/150 | 4/150 | 6/150 | 3/150 | 1/139 | 0/139
Other Adverse Events (participants affected / at risk) | 145/150 | 141/150 | 0/0 | 0/0 | 58/139 | 54/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC, MDV With Preservative: Infant Series (N=150) | 13vPnC, PFS Without Preservative: Infant Series (N=150) | 13vPnC, MDV: Between Infant Series and Toddler Dose (N=150) | 13vPnC, PFS: Between Infant Series and Toddler Dose (N=150) | 13vPnC, MDV With Preservative: Toddler Dose (N=139) | 13vPnC, PFS Without Preservative: Toddler Dose (N=139)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 4 | 2 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 2 | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC, MDV With Preservative: Infant Series (N=150) | 13vPnC, PFS Without Preservative: Infant Series (N=150) | 13vPnC, MDV: Between Infant Series and Toddler Dose (N=0) | 13vPnC, PFS: Between Infant Series and Toddler Dose (N=0) | 13vPnC, MDV With Preservative: Toddler Dose (N=139) | 13vPnC, PFS Without Preservative: Toddler Dose (N=139)
Injection site pain-1 (General disorders) | 44 | 46 | 0 | 0 | 0 | 0
Injection site pain-2 (General disorders) | 117 | 125 | 0 | 0 | 33 | 26
Injection site swelling (General disorders) | 17 | 16 | 0 | 0 | 0 | 0
Pyrexia-1 (General disorders) | 12 | 7 | 0 | 0 | 0 | 0
Pyrexia-2 (General disorders) | 37 | 32 | 0 | 0 | 0 | 0
Swelling (General disorders) | 64 | 70 | 0 | 0 | 12 | 16
Upper respiratory tract infection (Infections and infestations) | 16 | 10 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 92 | 107 | 0 | 0 | 20 | 22
Hypersomnia (Increased sleep) (Nervous system disorders) | 105 | 116 | 0 | 0 | 10 | 25
Irritability (Psychiatric disorders) | 114 | 117 | 0 | 0 | 32 | 31
Erythema (Redness) (Skin and subcutaneous tissue disorders) | 52 | 49 | 0 | 0 | 11 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT03548337/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT03548337/SAP_001.pdf